CLINICAL TRIAL: NCT05007938
Title: A Phase II, Single Arm, Study to Assess Befotertinib and Icotinib as First-Line Treatment in Patients With Locally Advanced or Metastatic NSCLC and Sensitising EGFR Mutation
Brief Title: Befotertinib and Icotinib in Treatment-naive Patients With Advanced EGFR-Mutant Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-BF-IV01
Record Dates: First submitted 2021-08-08; First posted 2021-08-17 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib + Befotertinib (Experimental): * Icotinib（125 mg orally, three times daily）
  * Befotertinib（25 mg orally, three times daily）
  Interventions: Drug: Icotinib; Drug: Befotertinib

INTERVENTIONS:
Drug: Icotinib — Icotinib is a EGFR ihibitior.
  Other Names: Conmana
Drug: Befotertinib — An orally available, irreversible, third-generation，mutant-selective epidermal growth factor receptor（EGFR）inhibitor. Befotertinib combine with icotinib means that both drugs will be given together until disease progression or meet the discontinuation criteria.
  Other Names: D-0316

SUMMARY:
This research study is studying a combination of two drugs as a possible treatment for Non-Small Cell Lung Cancer (NSCLC) with an EGFR mutation.

DETAILED DESCRIPTION:
This is a phase II, single-arm study assessing the safety and efficacy of befotertinib (25mg three times daily, orally）combining with icotinib (125mg three times daily, orally) in patients with locally advanced or metastatic NSCLC that is known to be EGFR sensitising mutation (EGFRm) positive, treatment-naive and eligible for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Pathologically confirmed adenocarcinoma of the lung, with locally advanced or metastatic disease and not amenable to curative surgery or radiotherapy (stage IIIB, IIIC or IV disease based on the eighth edition of the American Joint Committee on Cancer (AJCC) TNM classification). Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Patients must be treatment-naive for locally advanced or metastatic NSCLC systemic antitumor therapy. Prior adjuvant and neo-adjuvant therapy (except for EGFR-TKIs) is permitted if have been completed at least 6 months prior to initiation of disease progression.
* The tumour tissues harbour one of the two common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R),either alone or in combination with other EGFR mutations, excluding co-mutation of Ex19del and L858R,assessed by central laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Predicted survival ≥ 3 months.
* At least 1 measurable tumor lesion without radiotherapy as per RECIST v1.1.
* Agree to use effective contraception during the study period and for at least 3 months after completion of the study treatment.
* Provision of informed consent prior to any study procedure.

Exclusion Criteria:

* Combined with other malignancy(except for clinically cured in situ cervix carcinoma, basal cell or squamous epithelial skin cancer,thyroid papillary carcinoma).
* Prior treatment with any EGFR-TKIs.
* Prior treatment with any systemic antitumor therapy for locally advanced or metastatic NSCLC.
* Previous traditional chinese medicine with an antitumor indication within 2 weeks before the first dose of study drug.
* Previous major surgery within 4 weeks before the first dose of study drug,or planing to have major surgery during study.
* Symptoms or signs worsened within 2 weeks before the first dose of study drug.
* Any unresolved toxicities from prior treatment greater than NCI CTCAE v4.03 grade 2 or higher.
* Spinal cord compression,symptomatic or unstable central nervous system (CNS) metastases that require the use of steroids .Patients who have a stable CNS status for at least 4 weeks before treatment will be allowed to join the study.
* Any clinical evidence of serious or uncontrolled systemic disease,including uncontrolled hypertension after drug treatment,active bleeding diatheses, previous or present thrombus,uncontrolled cardiovascular and cerebrovascular diseases.
* Active infection including hepatitis B,hepatitis C,syphilis and human immunodeficiency virus (HIV).
* Mean resting corrected QT interval (QTcF) ≥450 msec,obtained from 3 ECGs or any clinically important abnormalities in rhythm,conduction, morphology of resting ECG or left ventricular ejection fraction (LVEF) ≤ 50%,etc.
* Previous history of interstitial lung disease(ILD),drug-induced interstitial lung disease,history of radiation-induced pneumonia requiring hormone therapy,or clinical evidence of active interstitial lung disease.
* Any instance that affects the patient's ability to swallow drug or oral malabsorption.
* Occur any laboratory indicator abnormalities as follow：

  * absolute neutrophil count(ANC)<1,500/mcL
  * platelets<100,000/mcL
  * hemoglobin<9.0 g/dL
  * AST/ALT>2.5 times the upper limit of normal (ULN)or >5 times the ULN in the presence of liver metastases
  * total bilirubin(TBIL)>1.5 times the ULN if no liver metastases or > 3 times the ULN in the presence of liver metastases
  * serum creatinine(SCr) >1.5 times the ULN or creatinine clearance ≥50 mL/min.
* Patients with a known allergy or delayed hypersensitivity reaction to the any component of study drugs or their excipients.
* Within 1 week before the first dose of study drug currently receiving or need concomitant medications known to be potent inhibitors or inducers of CYP3A, CYP2D6,CYPC8 and CYP2C19,sensitive substrate of CYP3A and CYP2C9.
* Within 1 week before the first dose of study drug ongoing use of warfarin.
* Previous therapeutic clinical trial within 4 weeks before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | 24 months
  ORR, per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of response（DOR） | 24 months
  DOR, defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death in the absence of disease progression.
Disease control rate（DCR） | 24 months
  DCR, defined as proportion of complete response, partial response, and disease stabilization to the proportion of patients with evalueable tumors.
Progression-free survival（PFS） | 36 months
  PFS, defined as time from study drug administration to progression or death due to any cause.
Intracranial objective response rate（iORR） | 24 months
  iORR, defined as the proportion of subjects with complete intracranial response, partial intracranial response to subjects with brain metastasis target lesions at baseline.
Overall survival （OS） | 36 months
  OS, defined as the time from study drug administration until the date of death due to any cause.
Adverse event（AE） | 36 months
  AE,defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study medication, whether or not considered related to the study drugs. AEs are summarized by type, incidence, severity and relationship to study drugs.

OTHER OUTCOMES:
AUC | 4 months
  AUC, defined as area under the plasma concentration-time curve.
Tmax | 4 months
  Tmax, defined as time of maximum concentration.
Cmax | 4 months
  Cmax,defined as maximum concentration.
Health Relevent Quality of Life（HRQoL） | 36 months
  Change from baseline scores on the functional assessment of cancer therapy- Lung (FACT-L) quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ye, MD, Principal Investigator — The First Affiliated Hospital of Xiamen University
Locations (1):
- Feng Ye, Xiamen, Fujian, China